CLINICAL TRIAL: NCT02166489
Title: Evaluation the Effect of Mesenchymal Stem Cells Transplantation in Patients With Chronic Renal Failure Due to Autosomal Dominant Polycystic Kidney Disease
Brief Title: Mesenchymal Stem Cells Transplantation in Patients With Chronic Renal Failure Due to Polycystic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Kidney-003
Record Dates: First submitted 2014-06-14; First posted 2014-06-18 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Renal Failure; Polycystic Kidney Disease
Keywords: autologous mesenchymal stem cells; polycystic kidney disease; intravenous injection; CRF
MeSH Terms: conditions — Kidney Failure, Chronic; Polycystic Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mesenchymal stem cell transplantation (Experimental): Intravenous injection of mesenchymal stem cell in patients with PKD
  Interventions: Biological: Intravenous injection autologous mesenchymal stem cells

INTERVENTIONS:
Biological: Intravenous injection autologous mesenchymal stem cells — Intravenous injection of mesenchymal stem cell in patients with PKD

SUMMARY:
This study was designed to provide confirmation of safety of mesenchymal stem cells (MSCs) therapy in chronic renal failure due to autosomal dominant polycystic kidney disease (ADPKD).

DETAILED DESCRIPTION:
The investigators will assess the 18-month safety and potential efficacy of autologous MSCs as therapy for ADPKD. A total of 6 patients with ADPKD IV injection of high doses 2×106 of autologous mesenchymal stem cells / kg their weight, which will be derived from biopsies of their bone marrow. Assessments will be made at 1, 3, 6, 12 and 18 months after cell injection. Changes in GFR rate were evaluated by scan isotope.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* ADPKD symptoms
* ADPKD confirmed with sonography and genetic testing
* Patient's age between 18 - 60 years
* GFR GFR 25-60 mL/min/1.73 m2
* Ability to understand and willingness to sign consent from

Exclusion Criteria:

* Pregnancy or breastfeeding
* Associated Cardiovascular disease
* Diabetes requiring medical intervention
* Other systemic diseases involving the kidneys, such as cancer, autoimmune diseases, blood diseases, liver disease, etc.
* Hospitalization due to illness in the last two months
* Life expectancy of less than two years
* Any allergies to the ingredients used in the cell culture

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mass formation | 1 month
  Evaluation the probability of mass formation in patients with PKD after mesenchyma l stem cell transplantation.

SECONDARY OUTCOMES:
Glomerular Filtration Rate (GFR) | 6 months
  Evaluation the acceleration of Glomerular Filtration Rate (GFR) in patients after mesenchymal stem cell transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Department of Regenerative Medicine & Cell therapy center of Royan Institute; Atieh Makhlough, MD, Study Director — Mazandaran University of Medical Sciences, Mazandaran, Iran.; Reza Moghadasali, PhD, Principal Investigator — Department of Regenerative Medicine And Royan Cell Therapy Center Royan Institute For stem Cell Biology and Technology
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Makhlough A, Shekarchian S, Moghadasali R, Einollahi B, Hosseini SE, Jaroughi N, Bolurieh T, Baharvand H, Aghdami N. Safety and tolerability of autologous bone marrow mesenchymal stromal cells in ADPKD patients. Stem Cell Res Ther. 2017 May 23;8(1):116. doi: 10.1186/s13287-017-0557-7. PMID 28535817
- See also: Related Info — http://Royaninstitute.org